CLINICAL TRIAL: NCT03469856
Title: ASET Clinical Investigational Plan Acetyl Salicylic Elimination Trial: The ASET Pilot Study
Brief Title: Acetyl Salicylic Elimination Trial: The ASET Pilot Study
Acronym: ASET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pedro A. Lemos (Other)
Collaborators: Imperial College London (Other); Cardialysis B.V. (Industry)
Responsible Party: Sponsor-Investigator, Pedro A. Lemos, MD, PhD, InCor Heart Institute
Organization: InCor Heart Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC 4579/17/079
Record Dates: First submitted 2018-02-21; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Monotherapy After PCI

STUDY DESIGN:
Intervention Model Description: The ASET Pilot study is a multicenter, single arm, open-label trial of single antiplatelet therapy with prasugrel for patients undergoing successful and optimal PCI for chronic stable angina with normal cardiac biomarkers values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): The ASET Pilot study is a multicenter, single arm, open-label trial of single antiplatelet therapy with prasugrel for patients undergoing successful and optimal PCI for chronic stable angina with normal cardiac biomarkers values. angiographic and/or findings from intracoronary imaging, only then patients will be enrolled in the study and loaded with prasugrel 60 mg and continued with prasugrel only (10 mg once a day) for three months. Aspirin and clopidogrel will be discontinued. At the 3-months follow-up visit, prasugrel (only) will be replaced by aspirin (only) or dual-antiplatelet therapy according to local standard of care.
  Interventions: Drug: Prasugrel monotherapy

INTERVENTIONS:
Drug: Prasugrel monotherapy — A multicenter, single arm, open-label trial of in patients with chronic stable angina
  Other Names: PCI with the SYNERGY® stent

SUMMARY:
A multicenter, single arm, open-label trial of prasugrel monotherapy after PCI with the new-generation thin-strut biodegradable polymer everolimus-eluting SYNERGY® stent in patients with chronic stable angina

DETAILED DESCRIPTION:
Single antiplatelet therapy with prasugrel is safe in selected patients undergoing successful PCI with the new generation biodegradable polymer everolimus-eluting SYNERGY® stent.

To assess in a proof-of-concept study the safety of single antiplatelet therapy with prasugrel after PCI with a new generation biodegradable polymer drug eluting stent in terms of ischemic and bleeding outcomes.

The ASET Pilot study is a multicenter, single arm, open-label trial of single antiplatelet therapy with prasugrel for patients undergoing successful and optimal PCI for chronic stable angina with normal cardiac biomarkers values. The patients will be loaded with standard dual antiplatelet therapy according to local practice (usually aspirin 300 mg and clopidogrel 600 mg, unless patient is on long-term therapy) at least 2 hours prior to the diagnostic catheterization or PCI procedure. After PCI, if the results are considered to be satisfactory by the operator based on clinical (e.g. clinical status, ECG, etc.), angiographic and/or findings from intracoronary imaging, only then patients will be enrolled in the study and loaded with prasugrel 60 mg and continued with prasugrel only (10 mg once a day) for three months. Aspirin and clopidogrel will be discontinued. At the 3-months follow-up visit, prasugrel (only) will be replaced by aspirin (only) or dual-antiplatelet therapy according to local standard of care. Clinical follow-up with office visit will be performed at 3 months and telephone contacts at 1, and 4 months (final follow-up). All events will be adjudicated by an independent clinical events committee (CEC).

An independent Data Safety and Monitoring Board (DSMB) will monitor the individual and collective safety of the patients in the study during enrolment phase and up to 3 months follow-up (primary endpoint).

The ASET study is a proof-of-concept pilot, feasibility and safety study designed as a single arm, open label trial with a stopping rule based on the occurrence of definite stent thrombosis. Based on previous pilot studies, 200 patients will be enrolled. The trial will be terminated if more than three (>3) patients experience definite stent thrombosis following index procedure till 4 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Successful PCI with optimal acute stent implantation results (based on local standard of care by angiography and/or findings from intracoronary imaging and on investigators' discretion) of one or more everolimus-eluting SYNERGY® stent(s). Typically, optimal acute coronary stenting result is a combination of successful stent implantation at the target lesion with absence of significant residual diameter stenosis (<20%), no edge dissection, no thrombus, no major side branch occlusion, "no-reflow", no major stent under-expansion or major stent incomplete apposition.

  2. Everolimus-eluting SYNERGY® stent implantation was performed to treat:
  1. patients with at least one stenosis (angiographic, visually determined de novo lesions with ≥50% DS) in at least one major epicardial territory (LAD and/or side branch, CX and/or side branch, RCA and/or side branch) with a vessel size between 2.25 mm and 4.0 mm in diameter supplying viable myocardium without left main stem involvement;
  2. Non-acute coronary disease, with normal cardiac troponin values prior to the PCI procedure, and evidences of myocardial ischemia by symptoms or non-invasive testing (e.g. treadmill exercise test, radionuclide scintigraphy, stress echocardiography);
  3. patients anatomical SYNTAX Score < 23 prior to everolimus-eluting SYNERGY® stent implantation; 3. Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site;

     Exclusion Criteria:
* Candidates will be ineligible for enrolment in the study if any of the following conditions apply:

  1. Under the age of 18 years or ≥ 75 years;
  2. Patients weighing < 60 kg;
  3. Unable to give Informed Consent;
  4. Females of child-bearing potential unless negative pregnancy test at screening and willing to use effective contraception (i.e. established use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or barrier methods of contraception with spermicide or sole male partner with prior vasectomy and confirmed absence of sperm in ejaculate) for the duration of treatment with study medication.
  5. Female who is breastfeeding at time of enrolment;
  6. Previous PCI in the last 12 months;
  7. Current (same hospitalization) or previous (within 12 months) acute coronary syndrome
  8. Patient with following lesion characteristics prior to everolimus-eluting SYNERGY® stent implantation:
* Left-main disease
* Chronic Total Occlusion
* Bifurcation lesion requiring two stent treatment
* Saphenous or arterial graft
* Severe calcification necessitating the use of rotablator 9. Patients with any previous history of definite stent thrombosis. 10. Patients treated with everolimus-eluting SYNERGY® stent(s) but who also concomitantly received any other non-study stent at the same procedure (all lesions must be treated with everolimus-eluting SYNERGY® stent); 11. Patients with planned PCI or surgical intervention to treat any cardiac or non-cardiac condition within the next 6 months; 12. Concomitant cardiac valve disease requiring surgical therapy (reconstruction or replacement); 13. Atrial fibrillation or other indication for oral anticoagulant therapy; 14. Known allergy to aspirin, prasugrel or diagnosed lactose intolerance; 15. Glomerular filtration rate below 60mL/min; 16. Previous stroke or transient ischemic cerebrovascular accident (TIA); 17. Previous history of intracranial haemorrhage or other intracranial pathology associated with increased bleeding risk; 18. Haemoglobin <10 g/dL or other evidence of active bleeding; 19. Peptic ulceration documented by endoscopy within the last 3 months unless healing proven by repeat endoscopy; 20. Any other condition deemed by the investigator to place the patient at excessive risk of bleeding with prasugrel; 21. Participation in another trial with an investigational drug or device; 22. Co-morbidity associated with life expectancy less than 1 year; 23. Assessment that the subject is not likely to comply with the study procedures or have complete follow-up; 24. Known drug or alcohol dependence within the past 12 months as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-07-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Primary Ischemic Endpoint | 3 months
  Composite of cardiac death, target-vessel myocardial infarction (spontaneous >48 hours) orn definite stent thrombosis
Primary Bleeding Endpoint | 3 months
  BARC 3 - 5 bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute - InCor, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kogame N, Guimaraes PO, Modolo R, De Martino F, Tinoco J, Ribeiro EE, Kawashima H, Ono M, Hara H, Wang R, Cavalcante R, Moulin B, Falcao BAA, Leite RS, de Almeida Sampaio FB, Morais GR, Meireles GC, Campos CM, Onuma Y, Serruys PW, Lemos PA. Aspirin-Free Prasugrel Monotherapy Following Coronary Artery Stenting in Patients With Stable CAD: The ASET Pilot Study. JACC Cardiovasc Interv. 2020 Oct 12;13(19):2251-2262. doi: 10.1016/j.jcin.2020.06.023. Epub 2020 Sep 16. PMID 32950419